CLINICAL TRIAL: NCT07102706
Title: A Phase I Monotherapy Study Assessing the Safety and Efficacy of GR1803, a BCMA×CD3 Bispecific Antibody, in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Phase I Trial of GR1803 Injection in Patients With RRMM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GR1803-001
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 0.02ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 1ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 10ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 30ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 90ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 180ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 240ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 300ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection
- 360ug/kg GR1803 (Experimental)
  Interventions: Drug: GR1803 injection

INTERVENTIONS:
Drug: GR1803 injection — weekly dose up to week 24 , biweekly dose from week 24 to week 36, and triweekly dose from week 36 to week 52

SUMMARY:
All subjects will receive GR1803 injection until intolerable toxicity or investigator-assessed disease progression occurs (except in cases of disease progression due to discontinuation of the drug as a result of an adverse event) or until the subject has been administered the drug for 52 weeks or until the subject withdraws consent or until the investigator determines that the subject needs to be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-2.
* ≥18 years of age.
* Multiple myeloma must be measurable by central laboratory assessment:

Serum monoclonal paraprotein (M-protein) level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or

Light chain multiple myeloma without measurable disease in the serum or the urine:

Serum immunoglobulin free light chain (FLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.

Exclusion Criteria:

* Prior treatment with any BCMA-targeted therapy.
* Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
* Plasma cell leukemia , Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloid light-chain amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
DLT | 52 weeks
  Dose Limited Toxicity

SECONDARY OUTCOMES:
ORR | 52 weeks
  Sum of the proportions of patients with proven strict complete remission (sCR), complete remission (CR), very good partial remission (VGPR) and partial remission (PR)
Progression-free survival (PFS) | 52 weeks
  Time from enrollment to tumor progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol